CLINICAL TRIAL: NCT00506259
Title: A Phase One Treatment Trial of the Circadian Sleep Disturbance in Smith-Magenis Syndrome (SMS)
Brief Title: Treatment Strategies for Children With Smith-Magenis Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 070076; 07-HG-0076
Record Dates: First submitted 2007-07-21; First posted 2007-07-25 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-05-22

CONDITIONS: Developmental Delay Disorders; Chromosome Deletion; Mental Retardation; Sleep Disorders, Circadian Rhythm; Self Injurious Behavior
Keywords: Deletion 17p11.2; Melatonin; Phototherapy; Behavioral Phenotype; Developmental Delay/MR; Smith-Magenis Syndrome; Sleep Disturbance; SMS; Sleep Disorder
MeSH Terms: conditions — Developmental Disabilities; Chromosome Deletion; Intellectual Disability; Sleep Disorders, Circadian Rhythm; Self-Injurious Behavior; Smith-Magenis Syndrome; Parasomnias; Sleep Wake Disorders | interventions — Phototherapy

INTERVENTIONS:
Drug: dTR Melatonin (NIH CC PDS)
Device: Phototherapy (Bright Light)
Drug: Melatonin CR

SUMMARY:
This study will examine the effect of bright light or melatonin treatment on sleep in children with Smith-Magenis syndrome (SMS), a genetic disorder characterized by certain physical, behavioral and developmental features. Patients have a disrupted sleep cycle involving early waking, frequent daytime napping and frequent nighttime awakenings. Melatonin is a hormone normally produced at night in healthy people. People with SMS produce high levels of melatonin during the daytime and very low levels at night. This may affect their behavior, mood, attention span and sleep patterns.

Healthy volunteers between 18 and 45 years of age and children with SMS who are between 3 and 16 years of age may be eligible for this study.

Healthy subjects are admitted to the NIH Clinical Center overnight. In the morning they take one dose of time-release melatonin and have blood and saliva samples collected hourly from 7:00 AM to 6:00 PM.

Children with SMS participate in a 2-part study, as follows:

Part 1 Inpatient Trial

Pre-trial at-home phase: During the month before NIH inpatient admission, participants do the following:

* Wear an actiwatch device or keep a daily sleep diary to monitor daytime alertness, mood shifts and sleep patterns.
* Complete a behavior assessment survey related to the child s behaviors and sleep patterns.
* Obtain frequent body temperature measurements.
* Collect several saliva samples over a 24-hour period.

NIH admission phase:

* Children are admitted to the NIH Clinical Center for 2-3 nights for bright light treatment. They remain in their rooms for alternating periods of exposure to standard dim room light and bright light, using a light box placed within 3 to 5 feet of the child. An electroencephalogram (EEG) with additional electrodes to track eye movements is used to monitor the child s attention. Between 8AM and 6PM serial blood samples are collected to measure melatonin levels. A parent rates the child s mood and behavior during the 2-day test period.
* Children are admitted to the NIH Clinical Center for 2-3 nights for melatonin treatment. They take a single dose of melatonin or placebo tablet at bedtime. During the daytime, EEG electrodes are placed to track eye movements. Between 7 PM and 7 AM serial blood samples are collected to measure melatonin levels. A parent rates the child s behavior and mood as described for the bright light study.
* Children may receive either or both of the bright light and melatonin treatments.

Part 2 Outpatient Trial

Children participate in a combined bright light with melatonin trial at home. They undergo the same procedures outlined in the pre-trial at-home phase of Part 1 (actiwatch, behavior assessments, body temperature measurements, saliva samples) over an 11-week period. If saliva samples cannot be collected for melatonin testing, 24-hour urine samples may be collected instead.

DETAILED DESCRIPTION:
Smith-Magenis syndrome (SMS) is a rare (1/25,000) clinically recognizable syndrome, characterized by the following features: a distinct pattern of minor craniofacial and skeletal anomalies, expressive speech/language delays, psychomotor and growth retardation, and a striking neurobehavioral phenotype. This phenotype includes stereotypies, self-injurious and aggressive behaviors, and a chronic sleep disorder associated with an inverted circadian melatonin rhythm. Sleep disturbances include daytime sleepiness, early sleep onset, and early morning awakening. Disturbed sleep is the strongest predictor of maladaptive behavior in children with SMS. Diminished nocturnal sleep is virtually universal in SMS, representing a major challenge to the patient and family. The majority (greater than 95%) of cases are due to interstitial deletion of 17p11.2; however, rare cases due to RAI1 gene mutations are also reported.

One of the likely contributing factors to these sleep disturbances is an inverse circadian pattern of the sleep-promoting hormone, melatonin. In SMS, plasma melatonin is high during the day and low at night, which is opposite the normal pattern. The underlying reason for this regular daytime melatonin secretory pattern is unknown. To our knowledge this pattern is distinctive to persons with SMS and not found elsewhere. SMS therefore offers a unique human syndrome for the study of melatonin function. At the present time, there is no effective treatment for sleep disturbances in SMS. Moreover, there are currently no controlled treatment trials underway in the U.S. with the specific goal of correcting the disturbed sleep pattern observed in this disease.

The aim of this Phase 1 treatment trial is to improve the quality of nocturnal sleep and decrease the need for daytime sleep by restoring a normal circadian pattern of melatonin levels in children with Smith-Magenis syndrome (SMS). We predict that the inverse pattern of release can be corrected by the combination of non-pharmacological suppression of daytime melatonin release and pharmacological replacement of nocturnal melatonin. Negative behaviors associated with accumulated sleep debt are expected to diminish as sleep quality improves.

Two treatment modalities will be evaluated alone and in combination: 1) light-induced suppression of daytime melatonin release and delay of nighttime sleep; and 2) pharmacological replacement of nocturnal melatonin. Melatonin levels measured in blood (Pre- vs. Post-treatment) will serve as the primary outcome parameter. A dTR-melatonin tablet developed by the Clinical Center Pharmaceutical Development Services (CC-PDS) will be used in this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

SMS subjects enrolled in protocol 01-HG-0109 will be invited to participate in this study. Protocol 01-HG-0109 has approximately 90 SMS subjects.

SMS inpatient admissions for the dTR-MT trial will be deferred until the BL study completes 10 SMS subjects who demonstrate expected SMS inverted diurnal MT profiles at baseline (T0).

SMS Subjects (N=12-15 per each treatment goal; 60 total enrollment):

* Male and female, childhood (average 5-16 years old; under age 5 years on case-by-case basis), all ethnicities with confirmed diagnosis of SMS (del 17p11.2). In some cases, molecular cytogenetic FISH screening (RAI1 FISH probe) may be required to confirm the SMS diagnosis prior to enrollment.
* Prepubertal (less than or equal to Tanner stage II).
* No history of seizures
* Priority will be given to subjects who are medication free and/or willing to discontinue sleep/behavioral medications during the study trial. We anticipate significant interest from families whose children are currently enrolled in the 01-HG-0109 protocol. We will also consider drug-free new referrals (self-referrals and/or via health care providers) eligible for enrollment.
* Documented sleep disturbance (by sleep log diary and/or actigraphy).

Unaffected Healthy Control Subjects (N=15). The pharmacokinetics of melatonin release by the dTR tablet will be evaluated in unaffected healthy control subjects prior to use in the inpatient SMS trial.

* Males and females of any ethnicity and between the ages 18-45 years.
* Regular (11PM - 7AM) sleep schedule for at least 1 week prior to study.
* Non-smokers, who have no history of seizures.
* Willing to discontinue coffee consumption for a period of 1-2 weeks prior to trial.
* BMI within normal limits (10-90 percentile).
* Unaffected with SMS.

EXCLUSION CRITERIA:

SMS Subjects:

* Inability to obtain informed consent.
* Failure to confirm clinical diagnosis of SMS by standard molecular cytogenetic (FISH) methods and/or DNA-based mutation analysis of RAI1 gene.
* Retinal diseases: macular degeneration, retinitis pigmentosa, diabetes, cataracts.
* Skin disease: Lupus (lupus erythematosis), history of skin cancer, history of adverse reaction(s) to sun (rash, reddening).
* Medications that are photosensitizing: Phenothiazines (Thorazine, Stelazine), Imipramine (AD), Porphyrins (antitumor), Chloroquine (antimalarial), Hydrocholorthiazine (antihypertensive, diuretic), Lithium (mood stabilizer) and/or antibiotics (Tetracycline).
* SMS subjects with extensive medication use may be excluded, depending on medications used and whether or not discontinuing medications for the trial presents a significant health risk. These include medications that might affect daytime vigilance (e.g., some seratonin antagonists such as Trazadone, SSRIs) and/or MAOIs, and/or antipsychotics (Risperidone), and/or some SSRIs (e.g., fluvoxamine) that affect the metabolism of melatonin and/or are strong CYP1A2 inhibitors.

Healthy Adult Controls:

* Individuals who have been diagnosed with a sleep disorder (e.g, restless legs, sleep apnea) known to impact sleep may be excluded at the discretion of the PI.
* Not willing to discontinue caffeine consumption (chocolate, coffee, tea) during study period.
* Persons with extensive medication use may be excluded, depending on medications used and whether or not discontinuing medications for the trial presents a significant health risk. These include medications that might affect daytime vigilance (e.g., some seratonin antagonists such as Trazadone, SSRIs) and/or MAOIs, and/or antipsychotics (Risperidone), and/or some SSRIs (e.g., fluvoxamine) that affect the metabolism of melatonin and/or are strong CYP1A2 inhibitors.
* Employed on a shift work schedule.
* Transmeridian travel within the last 2 weeks.
* Currently using melatonin.
* Women currently taking oral contraceptives (BCPs)
* Pregnant women and/or nursing mothers

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-07-17; Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Change in level of melatonin (pg/ml) from baseline

SECONDARY OUTCOMES:
Improved sleep parameters (actigraphy). Increased daytime vigilance. Decreased maladaptive behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bi W, Saifi GM, Shaw CJ, Walz K, Fonseca P, Wilson M, Potocki L, Lupski JR. Mutations of RAI1, a PHD-containing protein, in nondeletion patients with Smith-Magenis syndrome. Hum Genet. 2004 Nov;115(6):515-24. doi: 10.1007/s00439-004-1187-6. Epub 2004 Sep 30. PMID 15565467
- [Background] Slager RE, Newton TL, Vlangos CN, Finucane B, Elsea SH. Mutations in RAI1 associated with Smith-Magenis syndrome. Nat Genet. 2003 Apr;33(4):466-8. doi: 10.1038/ng1126. Epub 2003 Mar 24. PMID 12652298
- [Background] De Leersnyder H, De Blois MC, Claustrat B, Romana S, Albrecht U, Von Kleist-Retzow JC, Delobel B, Viot G, Lyonnet S, Vekemans M, Munnich A. Inversion of the circadian rhythm of melatonin in the Smith-Magenis syndrome. J Pediatr. 2001 Jul;139(1):111-6. doi: 10.1067/mpd.2001.115018. PMID 11445803